CLINICAL TRIAL: NCT05914649
Title: Neurocognitive Testing in Long COVID and Postural Tachycardia Syndrome Patients with Normal Saline: a Pilot Study
Brief Title: NC Testing in LC & POTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB23-0202
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Postural Orthostatic Tachycardia Syndrome; Post Acute Sequelae of SARS CoV 2 Infection
Keywords: POTS; Long COVID; Cognitive; Brain Fog
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Post-Acute COVID-19 Syndrome; Mental Fatigue | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will complete both the active and placebo arms of the study in a random order.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the person administering the cognitive testing will be blinded to the volume of saline infused (999 mL or 50 mL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 999 mL normal Saline (Experimental): 999 mL of normal saline infused intravenously.
  Interventions: Other: IV normal saline (999 mL infusion)
- 50 mL normal Saline (Placebo Comparator): 50 mL of normal saline infused intravenously.
  Interventions: Other: IV normal saline (50 mL infusion)

INTERVENTIONS:
Other: IV normal saline (999 mL infusion) — 999 mL of IV normal saline will be infused intravenously
  Arms: 999 mL normal Saline
Other: IV normal saline (50 mL infusion) — 50 mL of IV normal saline will be infused intravenously as a placebo control.
  Arms: 50 mL normal Saline

SUMMARY:
Patients with Postural Orthostatic Tachycardia Syndrome (POTS) and Post-Acute Sequelae of COVID (PASC, or "Long COVID") experience cognitive dysfunction. The investigators will test the hypothesis that 999 mL of IV saline will improve cognitive function in patients with POTS and Long COVID compared to placebo (50 mL of saline).

DETAILED DESCRIPTION:
Many POTS patients report cognitive dysfunction, otherwise referred to as brain fog, mental fog, mental clouding, or mental fatigue. Importantly, this cognitive dysfunction can occur even while lying down or seated, limiting the ability to engage in work and educational activities. Despite the prevalence and clinical impact of cognitive dysfunction in POTS, there are limited studies examining this phenomenon. Many patients with post-acute sequelae of SARS-COV-2 (PASC, or "Long COVID") experience symptoms such as subjective cognitive impairment ("brain fog"), fatigue, memory loss, headache, and fluctuation of blood pressure, amongst other signs and symptoms. Compared to healthy controls, this study will measure cognitive function in patients with POTS and Long COVID. This study will also evaluate IV normal saline (999 mL infusion) as a potential treatment for reduced cognitive function in POTS and Long COVID. This cross-over study will use a 50 mL saline infusion as a placebo control.

The findings from this study will be an initial first step towards understanding any neurocognitive impairment in participants with long COVID and POTS patients. This is a critical first step to future studies to assess underlying pathophysiology and potential treatments.

Primary hypothesis: Some objective measures of neurocognitive functions will improve in Long COVID and POTS patients after the infusion of 999 mL of normal saline compared to 50mL placebo control.

The primary analysis will compare the standing 5RTI task on the CANTAB testing scores between 999 mL saline infusion and 50 mL saline infusion (placebo).

Study Day and Instrumentation:

* A trained research staff member will insert an intravenous line in the vein of the participant's arm to administer either 999 mL or 50 mL of normal saline, which can take up to 30 minutes.
* After instrumentation, the participant will lie supine for at least 10 minutes while their ECG and BP are continuously recorded.
* The participant will stand up quickly (within several seconds) and then stand quietly for about 11 minutes while the recording continues. The lying-to-stand procedure will allow us to assess the hemodynamics of IST, POTS, and OH. A chair will be provided to the participant at any time they want to sit down during the test.
* After the stand test, the participant will be asked to do the Trail-Making Test (TMT) in the standing position. They will be asked to join numbers and letters in a circle. This test should not take more than approximately 10 minutes. A chair will be provided if they want to sit down at any time during the test.
* The participant will then be seated comfortably in a chair with their feet on the floor. They will be asked to do the Heart Counting Task (HCT) test. The participant will be asked to count their heartbeats without using their hands or other means to feel their pulse, which might affect their performance. This test will take approximately 10 minutes.
* The research team will then de-instrument the participant except for the Blood Pressure cuff on the arm. The team will continue to monitor the blood pressure throughout the study.
* Neuropsychological testing of the cognitive domains of memory, attention and executive function will be assessed using the Cambridge Neuropsychological Test Automated Battery (CANTAB) both seated and standing.
* The seated cognitive testing period will last approximately 60 minutes.
* The participant will be asked to stand unaided for up to 30 minutes and repeat portions of the CANTAB tests. Blood Pressure will be monitored throughout the stand test. A chair will be provided to the participant in case they would want to sit down.
* At the end of each stand test, the investigators will assess the patient's symptoms using the Vanderbilt Orthostatic Symptoms Score (VOSS). VOSS is a 9-item symptom rating, with each item scoring from 0 (absent) to 10 (worst) for a total score ranging from 0 to 90.
* The study will then be finished. The investigators will remove the recording patches and electrodes.
* The participant will then be booked for the second visit according to their convenience, where all the tests will be repeated, including IV insertion and infusion of normal saline, supine, and stand, and the cognitive tests (CANTAB, TMT, and HCT). Repeating these tests will help the research team assess whether the cognitive functions will improve for the Long COVID and POTS patients with blood volume expansion with the infusion of normal saline.

CANTAB Testing Protocol: CANTAB tests have demonstrated sensitivity to detecting changes in neuropsychological performance and include tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control. The subtests that will be used in this study for seated cognitive function are: Reaction Time Test (psychomotor Speed), Rapid Visual Information processing (Attention), Paired Associates Learning (Visual Episodic Memory), Spatial Span (Working memory), Verbal Recognition Memory (Verbal memory), Multitasking Test (Executive Function - Inhibition), Stocking of Cambridge (Executive Function - Planning) and the Emotional Bias Task (Emotion Processing). All tests are administered using a touchscreen tablet, and participants will respond to each test on-screen. Standardized written and audio instructions are given to participants through the software, and practice trials are completed before each test, reducing practice effects. Seated testing will be completed in approximately 60 minutes. The Reaction Time Test, Rapid Visual Processing and Multi Tasking tests will be repeated upon standing and will take approximately 30 minutes to complete.

After the in-lab portion of the study, participants will complete a series of validated questionnaires through a paper or RedCap secure web application for assessment of psychiatric symptoms. A unique URL link will be sent to the participants via Redcap Survey. These online surveys will take approximately 60 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Long COVID
* SARS-COV2 test positive
* Symptoms > 12 weeks post COVID
* Subjective complaint of 'brain fog" or cognitive dysfunction
* Patients with diagnosis of Postural Orthostatic Syndrome (POTS) from the Calgary Autonomic Investigation and Management Clinic
* Subjective complaint of 'brain fog" or cognitive impairment
* Healthy participants
* Without POTS or "brain fog"
* Age 18 to 60 years
* Female and Male
* Able to give an informed consent

Exclusion Criteria:

* Patients with overt causes for POTS (e.g., dehydration, prolonged bed rest)
* An inability to safely withdraw from medicine(s) that could make test interpretation difficult and impossible.
* Other factors which are in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule.
* Unable to give an informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
5RTI Reaction Time task (Standing) | During Procedure (3 hours)
  5RTI Reaction Time Score (Standing) after 999 mL IV saline compared to 5RTI score after 50 mL IV saline measured in milliseconds (ms). The minimum score is 100 ms and the maximum score is 5100 ms. A longer time is a worse outcome.

SECONDARY OUTCOMES:
Reaction Time Test (Psychomotor Speed) | During Procedure (3 hours)
  Reaction Time Test score after 1500mL IV saline compared to after 50mL IV saline measured in milliseconds. The minimum score is 100 ms and the maximum score is 5100 ms. A longer time is a worse outcome.
Paired Associates Learning (Visual Episodic Memory) | During Procedure (3 hours)
  Paired Associates Learning score after 999 mL IV saline compared to after 50 mL IV saline measured in arbitrary units. The minimum score is 0 and the maximum score is 70. A higher score is a worse outcome.
Verbal Recognition Memory (Verbal memory) | During Procedure (3 hours)
  Verbal Recognition Memory test score after 999 mL IV saline compared to after 50 mL IV saline. The range is 0-18. A higher score is a better outcome.
Multitasking Test (Executive Function - Inhibition) | During Procedure (3 hours)
  Multitasking Test Time after 999 mL IV saline compared to after 50 mL IV saline measured in ms. The range is 100 - 2000 ms. A longer time is a worse is a worse outcome.

OTHER OUTCOMES:
Sitting heart rate | During Procedure (10 minutes)
  Sitting heart rate after 999 mL IV saline compared to after 50 mL IV saline.
Standing heart rate | During Procedure (10 minutes)
  Standing heart rate after 999 mL IV saline compared to after 50 mL IV saline.

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No